CLINICAL TRIAL: NCT06360770
Title: Assessement of Microcirculation With NIRS Predicts Sepsis Development in Mechanically Ventilated Patients With Severe Covid-19 Pneumonia
Brief Title: Assessement of Microcirculation With NIRS Predicts Sepsis Development in Patients With Severe Covid-19 Pneumonia
Status: Completed | Type: Observational
Sponsor: General and Teaching Hospital Celje (Other)
Responsible Party: Principal Investigator, Matej Podbregar, ICU Director, General and Teaching Hospital Celje
Other Study IDs: NIRSCovidSBCelje
Record Dates: First submitted 2024-04-09; First posted 2024-04-11 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Sepsis
Keywords: sepsis; microcirculation; NIRS; SarsCov19
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sepsis and septic shock are among main causes of death in patients with severe Covid-19 pneumonia. A few factors are proven to predict sepsis in these patients. WIth near infrared spectroscopy it is possible to detect microcirculatory changes typical for sepsis early in the course of disease. The hypothesis that changes in tissue oxygene saturation during vasoocclusive test predict sepsis as well as mortality in mechancally ventilated patients withe severe Covid-19 pneumonia will be tested.

DETAILED DESCRIPTION:
At the moment the majority of ICU admissions in Slovenia are due to severe Covid19 pneumonia. Despite intensive supportive treatment the mortality of these patients is high, around 30%. The main reason for ICU admission is respiratory failure, these patients usually do not have multiorgan failure on admisssion. In the early phase of disease the inflamatory, endothelial and microcirculatory response is different than that in "classic" septic shock. One of the most common complications later in the course of severe Covid19 pneumonia is sepsis, which is defined as a life threatening syndrome with the failure of one or more organs due to disregulated inflamatory host response. This definition can be connected to the majority of patients who die.

It is not well known which factors predict sepsis development in patients with severe Covid19 pneumnia. In a laboratory mode the coagulation abnormality have been shown to be one of them. One of the earliest features of sepsis are microcirculation dysfunction and oxygene consumption abnormalities. Many studies have shown that with near infrared spectroscopy, we can reliably assess these abnormalities. With this method the tissue oxygene saturation can be measured. With vasoocclusive test the rate of tissue deoxygenation during stagnant ischemia and the rate of reoxygenation after flow release can be determined. It has been shown that the inclination of both curves decreases in sepsis. The measurements have also prognostic value.

With the clinical study we want to detect the microcirculatory abnormalities, typical for sepsis, early in the course, before the clinical and laboratory signs of multiorgan failure develop.

Aim of the study is to test hypotheis that NIRS measurements can predict sepsis development early and that machanically ventilated (due to Covid 19 pneumonia) patients with microcirculatory abnormalities have worse prognosis than those with preserved microcirculatory function.

ELIGIBILITY:
Inclusion Criteria:

* Severe respiratory failure due to Covid19 pneumonia
* Sedated, mechanically ventilated patient

Exclusion Criteria:

* Sepsis with multiorgan failure present on admisssion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with Covid19 pneumonia and need for ventilatory support (invasive mechanical ventilation) admitted to medical ICU of a regional general hospital.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
sepsis development | 2 months

SECONDARY OUTCOMES:
mortality | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- SB Celje, Celje, Slovenia

IPD SHARING:
Plan to Share IPD: No